CLINICAL TRIAL: NCT01213342
Title: Omega-3 Fatty Acid Supplementation and Dry Eye
Brief Title: Omega-3 Fatty Acid Supplements and Dry Eye
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Researchers left institution
Sponsor: Ohio State University (Other)
Collaborators: Nordic Naturals (Industry)
Responsible Party: Kelly K. Nichols, Principal Investigator/Associate Professor, The Ohio State University, College of Optometry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010H0014; NCT01131338 (obsolete NCT alias)
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: dry eye disease
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): This group will receive Omega-3 EFA supplements for 8 weeks. They will take 4 capsules/day.
  Interventions: Dietary Supplement: Omega-3 Fatty Acid
- Placebo Group (Placebo Comparator): This group will receive placebo supplements for 8 weeks. They will take 4 capsules a day.
  Interventions: Dietary Supplement: Soybean Soft Gels

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acid — Each patient will be instructed to take 4 soft gel capsules per day (2 with the morning meal and 2 with the evening meal). They will continue this regimen for 8 weeks. The total daily amount included in 4 soft gels includes:
  * EPA (Eicosapentaenoic Acid) 1300mg
  * DHA (Docosahexaenoic Acid) 900 mg
  * Other Omega-3's 360mg
  * Total Omega 3's 2560 mg
  Other Names: Fish Oil Soft Gels; ProOmega
  Arms: Treatment Group
Dietary Supplement: Soybean Soft Gels — Each patient will be instructed to take 4 soft gel capsules per day (2 with the morning meal and 2 with the evening meal. The main ingredient in the placebos is soybean oil (95.6%).
  Other Names: Placebo Soft Gels
  Arms: Placebo Group

SUMMARY:
Omega-3 fatty acids have been associated with a decline in inflammation. As dry eye disease is associated with inflammation of the ocular surface (DEWS report, Ocular Surface, 2007), the investigators hypothesize that the omega-3 fatty acid supplements used in this study will help to improve dry eye signs, such as eye surface irritation (staining) and tear film osmolarity, which is an overall measure of tear film stability and dry eye status. Further, the investigators hypothesize that dry eye symptoms, the end result of dry eye disease, such as discomfort and burning, will also improve with supplementation.

DETAILED DESCRIPTION:
Dry Eye is a disorder of the tear film due to tear deficiency or excessive tear evaporation which causes damage to the exposed ocular surface and is associated with symptoms of ocular discomfort. If left untreated, severe dry eyes can lead to desiccation of the corneal epithelium, increased discomfort and sometimes loss of vision. Abundant evidence from animal models and clinical evaluations confirm that inflammation is an integral part of all moderate and severe Dry Eye Disease (DED) states and is likely to be significant in the pathogenesis leading to the chronicity of DED. Omega-3 essential fatty acids (EFAs) have been shown to have anti-inflammatory effects and inhibit multiple aspects of inflammatory response.

DED is a common and growing problem as our population ages, causing chronic pain and visual disturbance that is not adequately treated with current approaches. If left untreated, severe dry eyes can lead to desiccation of the corneal epithelium, increased discomfort and sometimes loss of vision.The benefits are the possibility of alleviating or eliminating these symptoms of DED and the clinical data that will be gained on the safety and efficacy of omega-3s, which are already being marketed over-the-counter for the treatment of DED without any hard scientific data. The potential benefits of treatment outweigh the minimal risk of participation.

This study hopes to discover more about the efficacy and tolerability of omega-3 EFA's in the treatment of dry eye and ocular surface disease.

ELIGIBILITY:
Inclusion Criteria:

* Each qualified participant will have an eye doctor's diagnosis of dry eye disease.
* Answers to both questions: "How often do your eyes feel dry, how often do your eyes feel irritated" will either be "Often or Constant." (Schaumberg)
* ≥ 18 years of age
* The current use of artificial tears at least one time per week.
* Be willing/able to return for all study visits and to follow instructions from the study investigator and his/her staff.
* Stable dosage for one month time of all ocular medications and systemic medications (includes Restasis).
* Be able to swallow large, soft gels.

Exclusion Criteria:

* Patients who are allergic to ingredients of the treatment or placebo soft gels (fish, soybean oil, citrus).
* Current diagnosis of ocular infection (e.g. bacterial, viral or fungal).
* History of ocular herpetic keratitis.
* Past or current history of liver disease.
* Current use of blood thinners.
* Eye surgery (including cataract surgery) within 6 months prior to randomization.
* Previous LASIK surgery.
* Pregnant or nursing/lactating.
* Participation in a study of an investigational drug or device within the past 30 days.
* Cognitive or psychiatric deficit that precludes informed consent or ability to perform requirements of the investigation.
* Changes in ocular or systemic medications in the past 30 days.
* Contact lens wearers.
* Glaucoma diagnosis and/or use of glaucoma medications.
* Current use of punctual plugs.
* Current use of EPA/DHA supplements in excess of 1 gram/day.
* Use of ocular steroids currently or in the past 7 days.
* Patients planning on changing dosage of eye medications during the study.
* Patients who have an allergy to fluorescein.
* Patients who take aspirin daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) | Baseline, 4 weeks into treatment, 8 weeks into treatment
  Based on previous unpublished work by our group (and others), it is suggestive that a 10 unit change in OSDI score may be clinically meaningful. There currently is no accepted survey instrument to monitor change in DED clinical trials, although the OSDI has wide acceptance clinically. This study will help define what unit of change may be clinically and statistically acceptable for future trials.

SECONDARY OUTCOMES:
Changes in Osmolarity (TearLab) value | Baseline, 4 weeks, 12 weeks
  The TearLab also has limited use in DED clinical trials. Our best estimate of a clinically meaningful change is 7 mOsm/kg (reported dry eye, 315mOsm/kg - reported normal, 308 mOsm/kg). Again, as this has never been assessed, these results here are pilot in nature.
Changes in Staining scores | Baseline, 4 weeks, 8 weeks
  Changes in average staining scores (average of 5 corneal regions; 6 conjunctival regions) and sum staining scores will be evaluated.
Changes in Tear proteomics | Baseline, 4 weeks, 8 weeks
  This portion of the study is exploratory in nature. iTRAQ proteomics using mass spectrometry and RayBiotech quantibody microarrays will be used evaluate changes in inflammatory mediators for future biomarker search and pathway analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly K Nichols, OD, MPH, PhD, Principal Investigator — The Ohio State University College of Optometry
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

REFERENCES:
- [Background] Barabino S, Rolando M, Camicione P, Ravera G, Zanardi S, Giuffrida S, Calabria G. Systemic linoleic and gamma-linolenic acid therapy in dry eye syndrome with an inflammatory component. Cornea. 2003 Mar;22(2):97-101. doi: 10.1097/00003226-200303000-00002. PMID 12605039
- [Background] Macri A, Giuffrida S, Amico V, Iester M, Traverso CE. Effect of linoleic acid and gamma-linolenic acid on tear production, tear clearance and on the ocular surface after photorefractive keratectomy. Graefes Arch Clin Exp Ophthalmol. 2003 Jul;241(7):561-566. doi: 10.1007/s00417-003-0685-x. Epub 2003 May 27. PMID 12768289
- [Background] Roncone M, Bartlett H, Eperjesi F. Essential fatty acids for dry eye: A review. Cont Lens Anterior Eye. 2010 Apr;33(2):49-54; quiz 100. doi: 10.1016/j.clae.2009.11.002. Epub 2009 Dec 23. PMID 20031476
- [Background] Massi D, Franchi A, Alos L, Cook M, Di Palma S, Enguita AB, Ferrara G, Kazakov DV, Mentzel T, Michal M, Panelos J, Rodriguez-Peralto JL, Santucci M, Tragni G, Zioga A, Dei Tos AP. Primary cutaneous leiomyosarcoma: clinicopathological analysis of 36 cases. Histopathology. 2010 Jan;56(2):251-62. doi: 10.1111/j.1365-2559.2009.03471.x. PMID 20102404
- [Background] Miljanovic B, Trivedi KA, Dana MR, Gilbard JP, Buring JE, Schaumberg DA. Relation between dietary n-3 and n-6 fatty acids and clinically diagnosed dry eye syndrome in women. Am J Clin Nutr. 2005 Oct;82(4):887-93. doi: 10.1093/ajcn/82.4.887. PMID 16210721